CLINICAL TRIAL: NCT00420485
Title: A Phase I Open-label, Multi-center Dose-escalation Study to Determine the Maximum Tolerated Dose (MTD) and Dose Limiting Toxicity of Gimatecan Administered in Two Different Schedules in Adult Patients With Advanced Solid Tumors
Brief Title: Dose-escalation Study of Gimatecan Administered in Two Different Schedules in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBQ707A2101; NCT00462163 (obsolete NCT alias)
Record Dates: First submitted 2007-01-08; First posted 2007-01-11 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Solid Tumors
Keywords: Maximum Tolerated Dose; Solid Tumors; Dose Limiting Toxicity; Topoisomerase-1 Inhibitor
MeSH Terms: interventions — ST 1481

ARMS (2):
- Daily times five schedule (Experimental)
  Interventions: Drug: gimatecan
- Continuous schedule, twice daily (Experimental)
  Interventions: Drug: gimatecan

INTERVENTIONS:
Drug: gimatecan

SUMMARY:
This study will evaluate the Maximum Tolerated Dose and dose limiting toxicity of gimatecan administered orally in patients with advanced solid tumors

ELIGIBILITY:
Inclusion criteria:

* Advanced or metastatic cancer
* 18 years and above

Exclusion criteria:

* Previous treatment with 4 or more cycles of carboplatin;
* Previous treatment with 2 or more courses of nitrosourea or mitomycin;
* Previous radiation therapy greater than or equal to 25% of the hematopoietic reserve;
* Severe and/or uncontrolled medical conditions

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Presence of dose limiting toxicities in a 56-day treatment period | 56 days

SECONDARY OUTCOMES:
safety and tolerability assessed by adverse events, serious adverse events | 112 days
pharmacokinetics of gimatecan and its metabolites(s) | 91 days
response rate assessed by anti-tumor activity | 112 days
investigate tumor-specific mutations | 57 days
Evaluate activity signal for both dose schedules at MTD in ovarian, endometrial, and SCLC | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- Canada (2):
  - Novartis Investigative Site, Vancouver, British Columbia
  - MD Anderson Cancer Center - Orlando, Toronto, Ontario
- Novartis Investigative Site, Copenhagen, Denmark
- France (4):
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Toulouse
- Germany (2):
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Enschede, Netherlands
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Madrid, Spain